CLINICAL TRIAL: NCT05041738
Title: Comparative Evaluation of the Efficacy of Intraoral Cryotherapy Versus Intracanal Cryotherapy on Postoperative Pain in Lower Molar Teeth With Irreversible Pulpitis and Symptomatic Apical Periodontitis Randomized Clinical Trial
Brief Title: Comparative Evaluation of the Efficacy of Intraoral Cryotherapy Versus Intracanal Cryotherapy on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Toka Mohamed Ezzat Kamel Soliman, Principal investigator, Resident at faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO 3-3-5 8/9/2021
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral Cryotherapy (Experimental)
  Interventions: Procedure: Intraoral Cryotherapy
- Intracanal Cryotherapy (Active Comparator)
  Interventions: Procedure: Intracanal Cryotherapy

INTERVENTIONS:
Procedure: Intraoral Cryotherapy — small ice packs wrapped in sterile gauze placed in the mouth on the vestibular surface of the treated tooth
  Arms: Intraoral Cryotherapy
Procedure: Intracanal Cryotherapy — Intracanal cryotherapy technique using 2.5°C cold saline irrigation as final irrigant
  Arms: Intracanal Cryotherapy

SUMMARY:
The aim of this study is to clinically compare the efficacy of intraoral cryotherapy versus intracanal cryotherapy after single visit root canal therapy in lower molars with irreversible pulpitis and symptomatic apical periodontitis

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy patient (ASA I or II).

Mandibular first molar teeth with:

* Preoperative sharp pain and symptomatic apical periodontitis
* Absence or slight widening in the periodontal ligament (PDL).
* Vital response of pulp tissue to cold pulp tester (ethyl chloride spray) .
* Positive response to percussion test

Exclusion Criteria:

1. Medically compromised patients.
2. Pregnant women.
3. Patients reporting bruxism or clenching.
4. Patients allergic to ciprofloxacin or metronidazole.
5. Teeth associated with acute periapical abscess and/or swelling.
6. Greater than grade I mobility or pocket depth greater than 5mm.
7. Size of periapical radiolucency is greater than 8 mm.
8. No restorability: Hopeless tooth.
9. Immature teeth.
10. Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 20 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessed using Visual Analogue scale | 6 hours post treatment
  Intensity of pain after root canal treatment will be recorded by the patient where "0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain."
Postoperative pain assessed using Visual Analogue scale | 12 hours post treatment
  Intensity of pain after root canal treatment will be recorded by the patient where "0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain."
Postoperative pain assessed using Visual Analogue scale | 24 hours post treatment
  Intensity of pain after root canal treatment will be recorded by the patient where "0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain."

SECONDARY OUTCOMES:
Postoperative pain assessed using Visual Analogue scale | 48 hours post treatment
  Intensity of pain after root canal treatment will be recorded by the patient where "0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain."
Postoperative pain assessed using Visual Analogue scale | 72 hours post treatment
  Intensity of pain after root canal treatment will be recorded by the patient where "0= no pain, 1-3= mild pain, 4-6= moderate pain, 7-10= severe pain."

OTHER OUTCOMES:
Number of analgesics taken by the patient | Up to 72 hours
  Number of analgesics taken by the patient after endodontic treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fayyad DM, Abdelsalam N, Hashem N. Cryotherapy: A New Paradigm of Treatment in Endodontics. J Endod. 2020 Jul;46(7):936-942. doi: 10.1016/j.joen.2020.03.019. Epub 2020 May 6. PMID 32386857
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090